CLINICAL TRIAL: NCT03565900
Title: A Phase 3, Randomized, Double-blind, Active Comparator-controlled, Multicenter Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 in Recipients of Allogeneic Hematopoietic Stem Cell Transplant (PNEU-STEM)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 in Allogeneic Hematopoietic Stem Cell Transplant Recipients (V114-022/PNEU-STEM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-022; V114-022 (Other: Merck Protocol Number); 2018-000066-11 (EudraCT Number)
Record Dates: First submitted 2018-06-12; First posted 2018-06-21 (Actual); Results first posted 2022-10-20 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V114 on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants will have received HSCT 90 to 180 days prior to Day 1. Those who develop chronic graft-versus-host-disease (GVHD) during the first year after HSCT will receive V114 instead of PNEUMOVAX™23 as their fourth dose.
  Interventions: Biological: V114; Biological: PNEUMOVAX™23
- Prevnar 13™ (Active Comparator): Participants will receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants will have received HSCT 90 to 180 days prior to Day 1. Those who develop chronic GVHD during the first year after HSCT will receive Prevnar 13™ instead of PNEUMOVAX™23 as their fourth dose.
  Interventions: Biological: Prevnar 13™; Biological: PNEUMOVAX™23

INTERVENTIONS:
Biological: V114 — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F (2 mcg each), serotype 6B (4 mcg) and Merck Aluminum Phosphate Adjuvant (125 mcg) in each 0.5 mL dose.
  Other Names: VAXNEUVANCE™; Pneumococcal 15-Valent Conjugate Vaccine
  Arms: V114
Biological: Prevnar 13™ — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg) and 6B (4.4 mcg), and aluminum phosphate adjuvant (125 mcg aluminum) in each 0.5 ml dose
  Arms: Prevnar 13™
Biological: PNEUMOVAX™23 — 23-valent pneumococcal polysaccharide vaccine with serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, 33F (25 mcg each) in each 0.5 mL dose

SUMMARY:
The purpose of this study is to 1) evaluate the safety and tolerability, and immunogenicity of blinded V114 and Prevnar 13™ within each vaccination group, and 2) evaluate the safety and tolerability, and immunogenicity of PNEUMOVAX™23 (administered as open label, 12 months after allogeneic hematopoietic stem cell transplant [allo-HSCT] in participants who do not develop chronic graft-versus-host disease [GVHD]).

ELIGIBILITY:
Inclusion Criteria:

* Received a human leukocyte antigen (HLA) compatible donor including haploidentical and mismatched (related or unrelated) first allogeneic HSCT (i.e., bone marrow or peripheral blood stem cell) 90 to 180 days prior to randomization.
* Received the allogeneic HSCT for acute lymphoblastic leukemia (ALL) in first or second remission, acute myeloid leukemia (AML) in first or second remission, chronic myeloid leukemia (CML) in first chronic or accelerated phase, Hodgkin's lymphoma, non-Hodgkin's lymphoma, myelodysplastic syndrome (MDS), myelofibrosis and myeloproliferative diseases, and non-malignant disease such as aplastic anemia or sickle cell disease in participants ≥18 years of age and any non-malignant disease for participants 3 to <18 years of age.
* Life expectancy >12 months after allogeneic HSCT, according to investigator judgement.
* Clinically stable engraftment according to investigator judgment.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies: a) not a woman of childbearing potential (WOCBP) OR b) a WOCBP who agrees to use acceptable contraceptive methods during the treatment period and for at least 6 weeks after the last dose of study intervention.

Exclusion Criteria:

* Receipt of a previous allogeneic HSCT.
* Received allogeneic HSCT with ex-vivo graft manipulation, in vivo T cell depletion with alemtuzumab, or haploidentical allogeneic HSCT with high dose anti-thymocyte globulin.
* Received allogeneic HSCT for multiple myeloma or, for participants ≥18 years of age only, for any nonmalignant diseases except sickle cell disease and aplastic anemia.
* Persistent or relapsed primary disease after allogeneic HSCT.
* History of severe GVHD (Grade 3 or 4 GVHD) after allogeneic HSCT.
* Planned organ transplantation after allogeneic HSCT.
* History of culture-positive pneumococcal disease occurring after allogeneic HSCT.
* Known hypersensitivity to any component of pneumococcal polysaccharide vaccine, pneumococcal conjugate vaccine, or any diphtheria toxoid-containing vaccine.
* History of acquired immunodeficiency such as documented HIV infection, or anatomic asplenia.
* Coagulation disorder contraindicating intramuscular vaccinations.
* Severe hepatic impairment (defined as Child-Pugh Class C) at Screening.
* Serum aspartate transaminase (AST) or alanine transaminase (ALT) >6 × upper limit of normal (ULN) or serum total bilirubin >2.5 × ULN at Screening.
* A WOCBP who has a positive urine or serum pregnancy test before the 1st vaccination.
* Received chimeric antigen receptor T-cell (CAR-T) therapy or checkpoint inhibitor directed therapy (i.e., anti-Programmed Cell Death (PD)-1) after allogeneic HSCT.
* Received or planned to receive anti-Cluster of Differentiation (CD) 20 B-cell targeted therapy (e.g., rituximab) after allogeneic HSCT.
* Non-study pneumococcal vaccine administered after allogeneic HSCT, or is expected to receive non-study pneumococcal vaccine during participation in the study.
* Is currently participating or has participated in an interventional clinical study with an investigational compound/agent or device within 2 weeks of participating in this current study, or plans to receive any investigational compound/agent or device (in addition to existing therapy) within 2 weeks of any vaccination, that in the opinion of the investigator would interfere with the evaluation of the study objectives.
* Is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence as assessed by the study investigator.
* Has history or current evidence of any condition, therapy, laboratory test result abnormality, or other circumstance that might expose the participant to risk by participating in the study, confound the results of the study, or interfere with the participant's participation for the full duration of the study.
* Is or has an immediate family member who is investigational site or Sponsor staff directly involved with this study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (52):
- United States (13):
  - Stanford Health Care ( Site 0005), Palo Alto, California
  - Children's Hospital Colorado ( Site 0166), Aurora, Colorado
  - University of Florida ( Site 0011), Gainesville, Florida
  - University of Chicago ( Site 0016), Chicago, Illinois
  - Indiana Blood and Marrow Transplantation ( Site 0001), Indianapolis, Indiana
  - University of Kansas Medical Center ( Site 0007), Kansas City, Kansas
  - Johns Hopkins - University ( Site 0023), Baltimore, Maryland
  - Children's Mercy Hospital ( Site 0167), Kansas City, Missouri
  - Montefiore Einstein Center ( Site 0164), The Bronx, New York
  - Cincinnati Children's Hospital Medical Center ( Site 0010), Cincinnati, Ohio
  - Cleveland Clinic Foundation ( Site 0168), Cleveland, Ohio
  - Oregon Health & Science University ( Site 0018), Portland, Oregon
  - Baylor College of Medicine - Texas Children's Hospital ( Site 0165), Houston, Texas
- Australia (6):
  - St. Vincent's Hospital ( Site 0041), Sydney, New South Wales
  - The Children s Hospital at Westmead ( Site 0191), Westmead, New South Wales
  - Royal Adelaide Hospital ( Site 0040), Adelaide, South Australia
  - Austin Health-Austin Hospital ( Site 0038), Heidelberg, Victoria
  - The Alfred Hospital ( Site 0037), Melbourne, Victoria
  - Royal Melbourne Hospital ( Site 0039), Parkville, Victoria
- Belgium (5):
  - Cliniques Universitaires Saint-Luc ( Site 0122), Brussels, Bruxelles-Capitale, Region de
  - UZ Leuven ( Site 0119), Leuven, Vlaams-Brabant
  - AZ Sint Jan Brugge-Oostende ( Site 0118), Bruges, West-Vlaanderen
  - AZ Delta ( Site 0120), Roeselare, West-Vlaanderen
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman ( Site 0121), Liège
- Brazil (3):
  - Hospital Sao Rafael ( Site 0049), Salvador, Estado de Bahia
  - Santa Casa de Misericordia de Belo Horizonte ( Site 0050), Belo Horizonte, Minas Gerais
  - Instituto de Cancer e Transplante de Curitiba ICTR ( Site 0051), Curitiba, Paraná
- Canada (3):
  - Nova Scotia Health Authority QEII-HSC ( Site 0033), Halifax, Nova Scotia
  - Juravinski Cancer Centre ( Site 0032), Hamilton, Ontario
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0031), Montreal, Quebec
- Colombia (3):
  - Hospital Pablo Tobon Uribe ( Site 0077), Medellín, Antioquia
  - Fundacion Valle del Lili ( Site 0073), Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A ( Site 0075), Cali, Valle del Cauca Department
- France (6):
  - CHU de Nice ( Site 0084), Nice, Alpes-Maritimes
  - Hopital Jean Minjoz Besancon ( Site 0085), Besançon, Doubs
  - CHU de Grenoble Hopital Nord ( Site 0083), La Tronche, Isere
  - CHRU de Lille - Hopital Claude Huriez ( Site 0090), Lille, Nord
  - CHU Henri Mondor ( Site 0081), Créteil, Val-de-Marne
  - Hopital Saint-Antoine ( Site 0089), Paris
- Germany (3):
  - Universitaetsklinikum Koeln ( Site 0105), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf ( Site 0107), Düsseldorf, North Rhine-Westphalia
  - Universitaetsmedizin Mainz ( Site 0106), Mainz, Rhineland-Palatinate
- Mexico (7):
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez ( Site 0187), Monterrey, Nuevo León
  - Servicio de hematologia Universidad Autonoma de Nuevo Leon ( Site 0057), Monterrey, Nuevo León
  - Instituto Nacional de Pediatria ( Site 0062), Mexico City
  - Hospital Infantil de Mexico Federico Gomez ( Site 0061), Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 0058), Mexico City
  - Hospital Espanol ( Site 0059), México
  - Instituto Nacional de Cancerologia. ( Site 0060), México
- Sweden (3):
  - Karolinska Universitetssjukhuset ( Site 0143), Stockholm, Stockholms Lan [se-01]
  - Akademiska Sjukhuset ( Site 0144), Uppsala, Uppsala Lan [se-03]
  - Sahlgrenska Universitetssjukhuset ( Site 0145), Gothenburg, Vastra Gotalands Lan [se-14]

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Wilck M, Cornely OA, Cordonnier C, Velez JD, Ljungman P, Maertens J, Selleslag D, Mullane KM, Nabhan S, Chen Q, Dagan R, Richmond P, Daus C, Geddie K, Tamms G, Sterling T, Patel SM, Shekar T, Musey L, Buchwald UK; V114-022 (PNEU-STEM) Study Group. A Phase 3, Randomized, Double-Blind, Comparator-Controlled Study to Evaluate Safety, Tolerability, and Immunogenicity of V114, a 15-Valent Pneumococcal Conjugate Vaccine, in Allogeneic Hematopoietic Cell Transplant Recipients (PNEU-STEM). Clin Infect Dis. 2023 Oct 13;77(8):1102-1110. doi: 10.1093/cid/ciad349. PMID 37338158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited male and female participants at least 3 years of age who have received allogeneic hematopoietic stem cell transplant (allo-HSCT) 90 to 180 days prior to randomization.
Pre-assignment Details: 263 adult participants and 14 pediatric participants (3 to 18 years of age) were randomized in a 1:1 ratio to receive either V114 or Prevnar 13™ on Day 1.
Groups:
- V114: Participants received single 0.5 mL intramuscular (IM) injection of V114 on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants received HSCT 90 to 180 days prior to Day 1. Those who developed chronic graft-versus-host-disease (GVHD) during the first year after HSCT received V114 instead of PNEUMOVAX™23 as their fourth dose.
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants will have received HSCT 90 to 180 days prior to Day 1. Those who developed chronic GVHD during the first year after HSCT received Prevnar 13™ instead of PNEUMOVAX™23 as their fourth dose.
Period: Overall Study
Arm/Group | V114 | Prevnar 13™
Started | 139 | 138
Vaccination 1 With V114 or Prevnar 13™ (PCV) (Day 1) | 139 | 135
Vaccination 2 With PCV (Day 30) | 135 | 128
Vaccination 3 With PCV (Day 60) | 130 | 124
Vaccination 4 With PNEUMOVAX™23 (PPV23) (12 Months After Allo-HSCT, Without Chronic GVHD) | 89 | 75
Vaccination 4 With PCV (12 Months After Allo-HSCT, With Chronic GVHD) | 29 | 37
Completed | 115 | 111
Not Completed | 24 | 27
Not completed — Disposition Unknown | 4 | 1
Not completed — Withdrawal By Parent/Guardian | 0 | 1
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Randomized By Mistake | 0 | 2
Not completed — Physician Decision | 7 | 11
Not completed — Death | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | Prevnar 13™ | Total
Number analyzed (Participants) | 139 | 138 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (16.0) | 46.3 (18.3) | 47.1 (17.1)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 5 | 4 | 9
  Adolescents (12-17 years) | 3 | 2 | 5
  Adults (18-64 years) | 108 | 107 | 215
  From 65-84 years | 23 | 25 | 48
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 62 | 119
  Male | 82 | 76 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 29 | 59
  Not Hispanic or Latino | 104 | 104 | 208
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 122 | 115 | 237
  More than one race | 5 | 15 | 20
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adult Participants: Percentage of Participants With a Solicited Injection-site Adverse Event Following Any of the First 3 Doses With V114 or Prevnar 13™
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following any of the first 3 doses of V114 or Prevnar 13™, the percentage of adult participants with solicited injection-site AEs was assessed. The solicited injection-site AEs were erythema, pain, and swelling.
Time Frame: Up to 5 days after any of the Day 1, Day 30, or Day 60 vaccinations (V114 or Prevnar 13™)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- V114 (Adult): Adult participants received single 0.5 mL intramuscular (IM) injection of V114 on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants received HSCT 90 to 180 days prior to Day 1. Those who developed chronic graft-versus-host-disease (GVHD) during the first year after HSCT received V114 instead of PNEUMOVAX™23 as their fourth dose.
- Prevnar 13™ (Adult): Adult participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants will have received HSCT 90 to 180 days prior to Day 1. Those who developed chronic GVHD during the first year after HSCT received Prevnar 13™ instead of PNEUMOVAX™23 as their fourth dose.
Arm/Group | V114 (Adult) | Prevnar 13™ (Adult)
Number analyzed (Participants) | 131 | 129
Percentage of Participants
  Injection site erythema | 20.6 [14.0 to 28.6] | 14.0 [8.5 to 21.2]
  Injection site pain | 88.5 [81.8 to 93.4] | 74.4 [66.0 to 81.7]
  Injection site swelling | 32.1 [24.2 to 40.8] | 17.8 [11.7 to 25.5]

2. Primary Outcome: Pediatric Participants: Percentage of Participants With a Solicited Injection-site Adverse Event Following Any of the First 3 Doses With V114 or Prevnar 13™
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following any of the first 3 doses of V114 or Prevnar 13™, the percentage of pediatric participants with solicited injection-site AEs was assessed. The solicited injection-site AEs were erythema, induration, pain, and swelling.
Time Frame: Up to 14 days after any of the Day 1, Day 30, or Day 60 vaccinations (V114 or Prevnar 13™)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- V114 (Pediatric): Pediatric participants received single 0.5 mL intramuscular (IM) injection of V114 on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants received HSCT 90 to 180 days prior to Day 1. Those who developed chronic graft-versus-host-disease (GVHD) during the first year after HSCT received V114 instead of PNEUMOVAX™23 as their fourth dose.
- Prevnar 13™ (Pediatric): Pediatric participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants will have received HSCT 90 to 180 days prior to Day 1. Those who developed chronic GVHD during the first year after HSCT received Prevnar 13™ instead of PNEUMOVAX™23 as their fourth dose.
Arm/Group | V114 (Pediatric) | Prevnar 13™ (Pediatric)
Number analyzed (Participants) | 8 | 6
Percentage of Participants
  Injection site erythema | 0.0 [0.0 to 36.9] | 33.3 [4.3 to 77.7]
  Injection site induration | 12.5 [0.0 to 52.7] | 33.3 [4.3 to 77.0]
  Injection site pain | 75.0 [34.9 to 96.8] | 83.3 [35.9 to 99.6]
  Injection site swelling | 25.0 [3.2 to 65.1] | 50.0 [11.8 to 88.2]

3. Primary Outcome: Adult Participants: Percentage of Participants With a Solicited Systemic Adverse Event Following Any of the First 3 Doses With V114 or Prevnar 13™
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following any of the first 3 doses of V114 or Prevnar 13™, the percentage of adult participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were arthralgia, fatigue, headache, and myalgia.
Time Frame: Up to 14 days after any of the Day 1, Day 30, or Day 60 vaccinations (V114 or Prevnar 13™)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Adult) | Prevnar 13™ (Adult)
Number analyzed (Participants) | 131 | 129
Percentage of Participants
  Arthralgia | 16.0 [10.2 to 23.5] | 18.6 [12.3 to 26.4]
  Fatigue | 45.0 [36.3 to 54.0] | 40.3 [31.8 to 49.3]
  Headache | 29.0 [21.4 to 37.6] | 31.0 [23.2 to 39.7]
  Myalgia | 48.9 [40.0 to 57.7] | 34.9 [26.7 to 43.8]

4. Primary Outcome: Pediatric Participants: Percentage of Participants With a Solicited Systemic Adverse Event Following Any of the First 3 Doses With V114 or Prevnar 13™
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following any of the first 3 doses of V114 or Prevnar 13™, the percentage of pediatric participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were arthralgia, fatigue, headache, myalgia, and hives or welts.
Time Frame: Up to 14 days after any of the Day 1, Day 30, or Day 60 vaccinations (V114 or Prevnar 13™)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Pediatric) | Prevnar 13™ (Pediatric)
Number analyzed (Participants) | 8 | 6
Percentage of Participants
  Arthralgia | 12.5 [0.3 to 52.7] | 0.0 [0.0 to 45.9]
  Fatigue | 25.0 [3.2 to 65.1] | 16.7 [0.4 to 64.1]
  Headache | 12.5 [0.3 to 52.7] | 16.7 [0.4 to 64.1]
  Myalgia | 50.0 [15.7 to 84.3] | 16.7 [0.4 to 64.1]
  Hives or welts | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.

5. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event Up to Month 12 After Allogeneic HSCT
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. The percentage of participants with a vaccine-related SAE following dose 1 (with either V114 or Prevnar 13™) was reported. Vaccine-related SAEs were counted starting after vaccine dose 1 up to 12 months post-HSCT, which could be up to 9 months post-vaccine dose 1.
Time Frame: Up to 9 months
Population: All randomized participants who received at least 1 dose of the relevant study vaccination for the timepoint of interest were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Adult) | Prevnar 13™ (Adult) | V114 (Pediatric) | Prevnar 13™ (Pediatric)
Number analyzed (Participants) | 131 | 129 | 8 | 6
Percentage of Participants | 0.8 [0.0 to 4.2] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 45.9]

6. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Immunoglobulin G (IgG) at 30 Days Following Dose 3 With V114 or Prevnar 13™ (Day 90)
Description: The GMC of serotype-specific IgG for the serotypes contained in V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay.
Time Frame: Day 90 (30 days after the Day 60 vaccinations with V114 or Prevnar 13™)
Population: All randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity endpoint and who had sufficient data to perform the analyses were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 105 | 88
µg/mL
  Serotype 1 (Shared) | 2.97 [2.22 to 3.99] | 1.90 [1.34 to 2.69]
  Serotype 3 (Shared) | 0.80 [0.63 to 1.02] | 0.52 [0.38 to 0.71]
  Serotype 4 (Shared) | 1.61 [1.23 to 2.11] | 1.52 [1.04 to 2.20]
  Serotype 5 (Shared) | 2.85 [2.13 to 3.81] | 1.91 [1.32 to 2.77]
  Serotype 6A (Shared) | 3.40 [2.42 to 4.76] | 2.79 [1.78 to 4.38]
  Serotype 6B (Shared) | 3.49 [2.45 to 4.98] | 2.86 [1.82 to 4.49]
  Serotype 7F (Shared) | 3.20 [2.38 to 4.30] | 3.01 [2.07 to 4.36]
  Serotype 9V (Shared) | 2.56 [1.94 to 3.38] | 1.83 [1.26 to 2.65]
  Serotype 14 (Shared): number analyzed (Participants) | 105 | 87
  Serotype 14 (Shared) | 6.50 [4.94 to 8.57] | 4.61 [3.17 to 6.69]
  Serotype 18C (Shared) | 3.84 [2.83 to 5.22] | 2.58 [1.76 to 3.79]
  Serotype 19A (Shared) | 5.03 [3.88 to 6.53] | 4.31 [3.00 to 6.20]
  Serotype 19F (Shared) | 5.03 [3.72 to 6.79] | 3.67 [2.53 to 5.33]
  Serotype 23F (Shared) | 3.59 [2.64 to 4.88] | 2.62 [1.66 to 4.15]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 105 | 86
  Serotype 22F (Unique to V114) | 4.09 [3.02 to 5.54] | 0.15 [0.11 to 0.20]
  Serotype 33F (Unique to V114) | 3.40 [2.58 to 4.48] | 0.39 [0.29 to 0.53]

7. Secondary Outcome: Adult Participants: Percentage of Participants With a Solicited Injection-site Adverse Event Following Vaccination With PNEUMOVAX™23
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following a single dose vaccination with PNEUMOVAX™23, the percentage of adult participants with solicited injection-site AEs was assessed. The solicited injection-site AEs were erythema, pain, and swelling.
Time Frame: Up to 5 days after the PNEUMOVAX™23 vaccination (12 months after HSCT and approximately 6 to 9 months after Day 1)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Adult) | Prevnar 13™ (Adult)
Number analyzed (Participants) | 84 | 71
Percentage of Participants
  Injection site erythema | 17.9 [10.4 to 27.7] | 22.5 [13.5 to 34.0]
  Injection site pain | 67.9 [56.8 to 77.6] | 57.7 [45.4 to 69.4]
  Injection site swelling | 21.4 [13.2 to 31.7] | 23.9 [14.6 to 35.5]

8. Secondary Outcome: Pediatric Participants: Percentage of Participants With a Solicited Injection-site Adverse Event Following Vaccination With PNEUMOVAX™23
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following single dose vaccination with PNEUMOVAX™23, the percentage of pediatric participants with solicited injection-site AEs was assessed. The solicited injection-site AEs assessed were induration, pain, swelling, and erythema.
Time Frame: Up to 14 days after the PNEUMOVAX™23 vaccination (12 months after HSCT and approximately 6 to 9 months after Day 1)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Pediatric) | Prevnar 13™ (Pediatric)
Number analyzed (Participants) | 5 | 4
Percentage of Participants
  Injection site induration | 0.0 [0.0 to 52.2] | 25.0 [0.6 to 80.6]
  Injection site pain | 60.0 [14.7 to 94.7] | 50.0 [6.8 to 93.2]
  Injection site swelling | 20.0 [0.5 to 71.6] | 25.0 [0.6 to 80.6]
  Injection site erythema | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.

9. Secondary Outcome: Adult Participants: Percentage of Participants With a Solicited Systemic Adverse Event Following Vaccination With PNEUMOVAX™23
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following a single dose vaccination with PNEUMOVAX™23, the percentage of adult participants with solicited systemic AEs was assessed. The solicited systemic AEs were arthralgia, fatigue, headache, and myalgia.
Time Frame: Up to 14 days after the PNEUMOVAX™23 vaccination (12 months after HSCT and approximately 6 to 9 months after Day 1)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Adult) | Prevnar 13™ (Adult)
Number analyzed (Participants) | 84 | 71
Percentage of Participants
  Arthralgia | 7.1 [2.7 to 14.9] | 8.5 [3.2 to 17.5]
  Fatigue | 22.6 [14.2 to 33.0] | 16.9 [9.0 to 27.7]
  Headache | 21.4 [13.2 to 31.7] | 19.7 [11.2 to 30.9]
  Myalgia | 32.1 [22.4 to 43.2] | 26.8 [16.9 to 38.6]

10. Secondary Outcome: Pediatric Participants: Percentage of Participants With a Solicited Systemic Adverse Event Following Vaccination With PNEUMOVAX™23
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following a single dose vaccination with PNEUMOVAX™23, the percentage of pediatric participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were fatigue, headache, myalgia, hives or welts, and arthralgia.
Time Frame: Up to 14 days after the PNEUMOVAX™23 vaccination (12 months after HSCT and approximately 6 to 9 months after Day 1)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Pediatric) | Prevnar 13™ (Pediatric)
Number analyzed (Participants) | 5 | 4
Percentage of Participants
  Fatigue | 20.0 [0.5 to 71.6] | 0.0 [0.0 to 60.2]
  Headache | 20.0 [0.5 to 71.6] | 0.0 [0.0 to 60.2]
  Myalgia | 40.0 [5.3 to 85.3] | 0.0 [0.0 to 60.2]
  Hives or welts | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.
  Arthralgia | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.

11. Secondary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event Following Vaccination With PNEUMOVAX™23
Description: A SAE is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. The percentage of participants with a vaccine-related SAE following a single dose vaccination with PNEUMOVAX™23 was reported.
Time Frame: Up to 1 month after PNEUMOVAX™23 vaccination (12 months after HSCT and approximately 6 to 10 months after Day 1)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Adult) | Prevnar 13™ (Adult) | V114 (Pediatric) | Prevnar 13™ (Pediatric)
Number analyzed (Participants) | 84 | 71 | 5 | 4
Percentage of Participants | 1.2 [0.0 to 6.5] | 0.0 [0.0 to 5.1] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 60.2]

12. Secondary Outcome: Adult Participants With GVHD: Percentage of Participants With a Solicited Injection-site Adverse Event Following Dose 4 With V114 or Prevnar 13™
Description: This end point applies to adult participants who developed GVHD within 12 months of HSCT and received V114 or Prevnar 13™ as the fourth vaccination. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following dose 4 with V114 or Prevnar 13™, the percentage of adult participants with solicited injection-site AEs was assessed. The solicited injection-site AEs were erythema, pain, and swelling.
Time Frame: Up to 5 days after the fourth V114 or Prevnar 13™ vaccination (12 months after HSCT and approximately 6 to 9 months after Day 1)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Adult) | Prevnar 13™ (Adult)
Number analyzed (Participants) | 27 | 36
Percentage of Participants
  Injection site erythema | 3.7 [0.1 to 19.0] | 8.3 [1.8 to 22.5]
  Injection site pain | 77.8 [57.7 to 91.4] | 61.1 [43.5 to 76.9]
  Injection site swelling | 22.2 [8.6 to 42.3] | 13.9 [4.7 to 29.5]

13. Secondary Outcome: Pediatric Participants With GVHD: Percentage of Participants With a Solicited Injection-site Adverse Event Following Dose 4 With V114 or Prevnar 13™
Description: This end point applies to pediatric participants who developed GVHD within 12 months of HSCT and received V114 or Prevnar 13™ as the fourth vaccination dose. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following dose 4 with V114 or Prevnar 13™, the percentage of pediatric participants with solicited injection-site AEs was assessed. The solicited injection-site AE assessed were pain, erythema, swelling, and induration.
Time Frame: Up to 14 days after the fourth V114 or Prevnar 13™ vaccination (12 months after HSCT and approximately 6 to 9 months after Day 1)
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Pediatric) | Prevnar 13™ (Pediatric)
Number analyzed (Participants) | 2 | 1
Percentage of Participants
  Injection site pain | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5]
  Injection site erythema | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.
  Injection site swelling | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.
  Injection site induration | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.

14. Secondary Outcome: Adult Participants With GVHD: Percentage of Participants With a Solicited Systemic Adverse Event Following Dose 4 With V114 or Prevnar 13™
Description: This end point applies to adult participants who developed GVHD within 12 months of HSCT and received V114 or Prevnar 13™ as the fourth vaccination dose. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following dose 4 with V114 or Prevnar 13™, the percentage of adult participants with solicited systemic AEs was assessed. The solicited systemic AEs were arthralgia, fatigue, headache, and myalgia.
Time Frame: as for outcome 13
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Adult) | Prevnar 13™ (Adult)
Number analyzed (Participants) | 27 | 36
Percentage of Participants
  Arthralgia | 11.1 [2.4 to 29.2] | 8.3 [1.8 to 22.5]
  Fatigue | 29.6 [13.8 to 50.2] | 16.7 [6.4 to 32.8]
  Headache | 22.2 [8.6 to 42.3] | 11.1 [3.1 to 26.1]
  Myalgia | 29.6 [13.8 to 50.2] | 22.2 [10.1 to 39.2]

15. Secondary Outcome: Pediatric Participants With GVHD: Percentage of Participants With a Solicited Systemic Adverse Event Following Dose 4 With V114 or Prevnar 13™
Description: This end point applies to pediatric participants who developed GVHD within 12 months of HSCT and received V114 or Prevnar 13™ as the fourth vaccination. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following dose 4 with V114 or Prevnar 13™, the percentage of pediatric participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed myalgia, arthralgia, headache, fatigue, and hives or welts.
Time Frame: as for outcome 13
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Pediatric) | Prevnar 13™ (Pediatric)
Number analyzed (Participants) | 2 | 1
Percentage of Participants
  Myalgia | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.
  Arthralgia | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.
  Headache | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.
  Fatigue | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.
  Hives or welts | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed. | 0.0 [NA to NA] — 95% Confidence Interval could not be calculated, because 0 events were observed.

16. Secondary Outcome: Participants With GVHD: Percentage of Participants With a Vaccine-related Serious Adverse Event Following Dose 4 With V114 or Prevnar 13™
Description: This end point applies to participants who developed GVHD within 12 months of HSCT and received V114 or Prevnar 13™ as vaccine dose 4. An SAE is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. The percentage of participants with a vaccine-related SAE following dose 4 with V114 or Prevnar 13™ through completion of study was reported.
Time Frame: Up to 6 months after the fourth V114 or Prevnar 13™ vaccination (12 months after HSCT and approximately 6 to 15 months after Day 1)
Population: All randomized participants who received at least 1 dose of relevant study vaccination for the timepoint of interest were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 (Adult) | Prevnar 13™ (Adult) | V114 (Pediatric) | Prevnar 13™ (Pediatric)
Number analyzed (Participants) | 27 | 36 | 2 | 1
Percentage of Participants | 0.0 [0.0 to 12.8] | 0.0 [0.0 to 9.7] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 97.5]

17. Secondary Outcome: Geometric Mean Titer of Serotype-specific Opsonophagocytic Activity at 30 Days Following Dose 3 With V114 or Prevnar 13™ (Day 90)
Description: The GMT of serotype-specific OPA for the serotypes contained in V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using a multiplexed opsonophagocytic assay.
Time Frame: Up to Day 90 (30 days after the Day 60 vaccinations with V114 or Prevnar 13™)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 92 | 68
Titers
  Serotype 1 (Shared) | 90.9 [60.8 to 135.9] | 59.3 [37.8 to 93.1]
  Serotype 3 (Shared): number analyzed (Participants) | 92 | 67
  Serotype 3 (Shared) | 152.1 [114.6 to 201.7] | 128.5 [89.6 to 184.4]
  Serotype 4 (Shared) | 1008.4 [684.3 to 1486.2] | 1357.7 [786.7 to 2343.1]
  Serotype 5 (Shared) | 317.6 [206.7 to 487.9] | 169.1 [106.1 to 269.6]
  Serotype 6A (Shared): number analyzed (Participants) | 91 | 68
  Serotype 6A (Shared) | 2494.5 [1731.4 to 3593.8] | 2295.0 [1463.8 to 3598.4]
  Serotype 6B (Shared): number analyzed (Participants) | 90 | 68
  Serotype 6B (Shared) | 2280.2 [1500.8 to 3464.3] | 3000.4 [1800.0 to 5001.3]
  Serotype 7F (Shared) | 1945.3 [1278.5 to 2960.0] | 3076.9 [1958.1 to 4834.7]
  Serotype 9V (Shared): number analyzed (Participants) | 92 | 66
  Serotype 9V (Shared) | 1059.4 [743.0 to 1510.5] | 1050.0 [659.5 to 1671.6]
  Serotype 14 (Shared): number analyzed (Participants) | 91 | 68
  Serotype 14 (Shared) | 1953.6 [1296.9 to 2942.9] | 1689.2 [995.0 to 2867.6]
  Serotype 18C (Shared): number analyzed (Participants) | 92 | 67
  Serotype 18C (Shared) | 1146.6 [833.6 to 1577.2] | 714.6 [439.3 to 1162.3]
  Serotype 19A (Shared) | 1365.6 [960.4 to 1941.8] | 1201.6 [724.0 to 1994.2]
  Serotype 19F (Shared): number analyzed (Participants) | 92 | 67
  Serotype 19F (Shared) | 965.6 [675.3 to 1380.8] | 1065.6 [707.8 to 1604.3]
  Serotype 23F (Shared): number analyzed (Participants) | 91 | 65
  Serotype 23F (Shared) | 1158.3 [784.1 to 1711.1] | 2065.2 [1144.3 to 3727.4]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 89 | 67
  Serotype 22F (Unique to V114) | 1127.5 [717.9 to 1770.7] | 19.0 [11.9 to 30.2]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 91 | 68
  Serotype 33F (Unique to V114) | 4441.7 [2966.6 to 6650.2] | 173.6 [97.0 to 310.7]

18. Secondary Outcome: Percentage of Participants With Geometric Mean Fold Rises (GMFR) ≥4 in Serotype-specific IgG at 30 Days Following Dose 3 With V114 or Prevnar 13™ (Day 90)
Description: The GMFR of serotype-specific IgG for the serotypes contained in V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay.
Time Frame: Day 1 (Baseline) and Day 90 (30 days after the Day 60 vaccinations with V114 or Prevnar 13™)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 103 | 84
Percentage of Participants
  Serotype 1 (Shared) | 69.9 [60.1 to 78.5] | 64.3 [53.1 to 74.4]
  Serotype 3 (Shared) | 62.1 [52.0 to 71.5] | 48.8 [37.7 to 60.0]
  Serotype 4 (Shared) | 73.8 [64.2 to 82.0] | 70.2 [59.3 to 79.7]
  Serotype 5 (Shared) | 60.2 [50.1 to 69.7] | 60.7 [49.5 to 71.2]
  Serotype 6A (Shared) | 73.8 [64.2 to 82.0] | 69.0 [58.0 to 78.7]
  Serotype 6B (Shared) | 71.8 [62.1 to 80.3] | 69.0 [58.0 to 78.7]
  Serotype 7F (Shared) | 69.9 [60.1 to 78.5] | 70.2 [59.3 to 79.7]
  Serotype 9V (Shared) | 65.0 [55.0 to 74.2] | 63.1 [51.9 to 73.4]
  Serotype 14 (Shared): number analyzed (Participants) | 103 | 83
  Serotype 14 (Shared) | 51.5 [41.4 to 61.4] | 50.6 [39.4 to 61.8]
  Serotype 18C (Shared) | 67.0 [57.0 to 75.9] | 61.9 [50.7 to 72.3]
  Serotype 19A (Shared) | 55.3 [45.2 to 65.1] | 48.8 [37.7 to 60.0]
  Serotype 19F (Shared) | 63.1 [53.0 to 72.4] | 61.9 [50.7 to 72.3]
  Serotype 23F (Shared) | 61.2 [51.1 to 70.6] | 61.9 [50.7 to 72.3]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 103 | 83
  Serotype 22F (Unique to V114) | 74.8 [65.2 to 82.8] | 1.2 [0.0 to 6.5]
  Serotype 33F (Unique to V114) | 54.4 [44.3 to 64.2] | 4.8 [1.3 to 11.7]

19. Secondary Outcome: Percentage of Participants With GMFR ≥4 in Serotype-specific OPA at 30 Days Following Dose 3 With V114 or Prevnar 13™ (Day 90)
Description: Activity for the 15 serotypes contained in V114 vaccine were determined using a Multiplex Opsonophagocytic Assay. The GMFR of serotype-specific OPA for the serotypes contained in V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using multiplexed opsonophagocytic assay.
Time Frame: Time Frame: Day 1 (Baseline) and Day 90 (30 days after the Day 60 vaccinations with V114 or Prevnar 13™)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 88 | 62
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 88 | 61
  Serotype 1 (Shared) | 65.9 [55.0 to 75.7] | 54.1 [40.8 to 66.9]
  Serotype 3 (Shared): number analyzed (Participants) | 88 | 61
  Serotype 3 (Shared) | 58.0 [47.0 to 68.4] | 55.7 [42.4 to 68.5]
  Serotype 4 (Shared): number analyzed (Participants) | 87 | 59
  Serotype 4 (Shared) | 71.3 [60.6 to 80.5] | 78.0 [65.3 to 87.7]
  Serotype 5 (Shared) | 70.5 [59.8 to 79.7] | 53.2 [40.1 to 66.0]
  Serotype 6A (Shared): number analyzed (Participants) | 87 | 61
  Serotype 6A (Shared) | 64.4 [53.4 to 74.4] | 68.9 [55.7 to 80.1]
  Serotype 6B (Shared): number analyzed (Participants) | 85 | 60
  Serotype 6B (Shared) | 69.4 [58.5 to 79.0] | 73.3 [60.3 to 83.9]
  Serotype 7F (Shared): number analyzed (Participants) | 86 | 60
  Serotype 7F (Shared) | 68.6 [57.7 to 78.2] | 71.7 [58.6 to 82.5]
  Serotype 9V (Shared): number analyzed (Participants) | 88 | 60
  Serotype 9V (Shared) | 54.5 [43.6 to 65.2] | 53.3 [40.0 to 66.3]
  Serotype 14 (Shared): number analyzed (Participants) | 86 | 62
  Serotype 14 (Shared) | 54.7 [43.5 to 65.4] | 58.1 [44.8 to 70.5]
  Serotype 18C (Shared): number analyzed (Participants) | 88 | 60
  Serotype 18C (Shared) | 69.3 [58.6 to 78.7] | 46.7 [33.7 to 60.0]
  Serotype 19A (Shared): number analyzed (Participants) | 86 | 61
  Serotype 19A (Shared) | 64.0 [52.9 to 74.0] | 59.0 [45.7 to 71.7]
  Serotype 19F (Shared): number analyzed (Participants) | 88 | 61
  Serotype 19F (Shared) | 61.4 [50.4 to 71.6] | 68.9 [55.7 to 80.1]
  Serotype 23F (Shared): number analyzed (Participants) | 85 | 55
  Serotype 23F (Shared) | 63.5 [52.4 to 73.7] | 69.1 [55.2 to 80.9]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 84 | 58
  Serotype 22F (Unique to V114) | 70.2 [59.3 to 79.7] | 3.4 [0.4 to 11.9]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 86 | 62
  Serotype 33F (Unique to V114) | 61.6 [50.5 to 71.9] | 11.3 [4.7 to 21.9]

ADVERSE EVENTS:
Time Frame: Non-serious AEs: Up to 14 days after each vaccination; SAEs and deaths (all-causes): Through 6 months after dose 4 with V114 or Prevnar13™ (up to 15 months total) or through 1 month after single dose vaccination with PNEUMOVAX™23 (up to 10 months total).
Description: The analysis population for deaths (all-causes) included all randomized participants. The analysis population for AEs included all randomized participants who received at least 1 dose of study vaccination.
Groups:
- V114 (Following Any of the First 3 Doses of PCV) Adults; V114 (Following PPV23) Adults; V114 (Following Dose 4 of PCV) Adults: Adult participants received single 0.5 mL intramuscular (IM) injection of V114 on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants received HSCT 90 to 180 days prior to Day 1. Those who developed chronic graft-versus-host-disease (GVHD) during the first year after HSCT received V114 instead of PNEUMOVAX™23 as their fourth dose.
- Prevnar 13™ (Following Any of the First 3 Doses of PCV) Adults; Prevnar 13™ (Following PPV23) Adults; Prevnar 13™ (Following Dose 4 of PCV) Adults: Adult participants received a single 0.5 mL intramuscular (IM) injection of Prevnar 13™ on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants will have received HSCT 90 to 180 days prior to Day 1. Those who developed chronic GVHD during the first year after HSCT received Prevnar 13™ instead of PNEUMOVAX™23 as their fourth dose.
- V114 (Following Any of the First 3 Doses of PCV) Pediatric; V114 (Following PPV23) Pediatric; V114 (Following Dose 4 of PCV) Pediatric: Pediatric participants received single 0.5 mL intramuscular (IM) injection of V114 on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants received HSCT 90 to 180 days prior to Day 1. Those who developed chronic graft-versus-host-disease (GVHD) during the first year after HSCT received V114 instead of PNEUMOVAX™23 as their fourth dose.
- Prevnar 13™ (Following Any of the First 3 Doses of PCV) Pediatric; Prevnar 13™ (Following PPV23) Pediatric; Prevnar 13™ (Following Dose 4 of PCV) Pediatric: Pediatric participants received a single 0.5 mL intramuscular (IM) injection of Prevnar 13™ on Day 1, Day 30 and Day 60 and a single 0.5 mL IM injection of PNEUMOVAX™23 at 12 months after HSCT. Participants will have received HSCT 90 to 180 days prior to Day 1. Those who developed chronic GVHD during the first year after HSCT received Prevnar 13™ instead of PNEUMOVAX™23 as their fourth dose.
Arm/Group | V114 (Following Any of the First 3 Doses of PCV) Adults | Prevnar 13™ (Following Any of the First 3 Doses of PCV) Adults | V114 (Following PPV23) Adults | Prevnar 13™ (Following PPV23) Adults | V114 (Following Dose 4 of PCV) Adults | Prevnar 13™ (Following Dose 4 of PCV) Adults | V114 (Following Any of the First 3 Doses of PCV) Pediatric | Prevnar 13™ (Following Any of the First 3 Doses of PCV) Pediatric | V114 (Following PPV23) Pediatric | Prevnar 13™ (Following PPV23) Pediatric | V114 (Following Dose 4 of PCV) Pediatric | Prevnar 13™ (Following Dose 4 of PCV) Pediatric
All-Cause Mortality (participants affected / at risk) | 6/131 | 9/129 | 1/84 | 0/71 | 2/27 | 1/36 | 1/8 | 0/6 | 0/5 | 0/4 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 38/131 | 48/129 | 2/84 | 4/71 | 6/27 | 7/36 | 2/8 | 1/6 | 0/5 | 0/4 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 125/131 | 108/129 | 65/84 | 53/71 | 22/27 | 26/36 | 7/8 | 6/6 | 3/5 | 3/4 | 1/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (Following Any of the First 3 Doses of PCV) Adults (N=131) | Prevnar 13™ (Following Any of the First 3 Doses of PCV) Adults (N=129) | V114 (Following PPV23) Adults (N=84) | Prevnar 13™ (Following PPV23) Adults (N=71) | V114 (Following Dose 4 of PCV) Adults (N=27) | Prevnar 13™ (Following Dose 4 of PCV) Adults (N=36) | V114 (Following Any of the First 3 Doses of PCV) Pediatric (N=8) | Prevnar 13™ (Following Any of the First 3 Doses of PCV) Pediatric (N=6) | V114 (Following PPV23) Pediatric (N=5) | Prevnar 13™ (Following PPV23) Pediatric (N=4) | V114 (Following Dose 4 of PCV) Pediatric (N=2) | Prevnar 13™ (Following Dose 4 of PCV) Pediatric (N=1)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyserositis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic graft versus host disease (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease (Immune system disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease in lung (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocardia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 6 (9) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion microchimerism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (Following Any of the First 3 Doses of PCV) Adults (N=131) | Prevnar 13™ (Following Any of the First 3 Doses of PCV) Adults (N=129) | V114 (Following PPV23) Adults (N=84) | Prevnar 13™ (Following PPV23) Adults (N=71) | V114 (Following Dose 4 of PCV) Adults (N=27) | Prevnar 13™ (Following Dose 4 of PCV) Adults (N=36) | V114 (Following Any of the First 3 Doses of PCV) Pediatric (N=8) | Prevnar 13™ (Following Any of the First 3 Doses of PCV) Pediatric (N=6) | V114 (Following PPV23) Pediatric (N=5) | Prevnar 13™ (Following PPV23) Pediatric (N=4) | V114 (Following Dose 4 of PCV) Pediatric (N=2) | Prevnar 13™ (Following Dose 4 of PCV) Pediatric (N=1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (15) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 59 (105) | 52 (111) | 19 (21) | 12 (16) | 8 (9) | 6 (6) | 2 (5) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 27 (37) | 18 (22) | 15 (15) | 16 (16) | 1 (1) | 3 (3) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 116 (284) | 97 (237) | 57 (57) | 41 (42) | 21 (21) | 22 (23) | 6 (13) | 5 (8) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 42 (64) | 23 (35) | 18 (18) | 17 (17) | 6 (7) | 5 (5) | 2 (3) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic graft versus host disease in skin (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Graft versus host disease in eye (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (33) | 24 (38) | 6 (6) | 6 (6) | 3 (3) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 64 (111) | 45 (77) | 27 (30) | 19 (20) | 8 (8) | 8 (8) | 4 (8) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 38 (73) | 40 (67) | 18 (20) | 14 (16) | 6 (7) | 4 (4) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT03565900/Prot_SAP_000.pdf